CLINICAL TRIAL: NCT06579885
Title: Mapping the Burden of Ocular Complications of Mpox in the Democratic Republic Congo (DRC)
Brief Title: Ocular Complications of Mpox in the Democratic Republic Congo
Acronym: MPOX-EYE
Status: Recruiting | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other)
Responsible Party: Sponsor
Other Study IDs: MPOX-EYE
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Monkeypox; Mpox (Monkeypox)
Keywords: ophthalmology; complications
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tear fluid samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study in which patients diagnosed with mpox will be enrolled, will undergo standard ophthalmological examinations of their eyes to see if there are any complications of mpox. The study will primarily assess the presence of ophthalmological signs and symptoms at enrollment.

DETAILED DESCRIPTION:
This is an observational study in which patients diagnosed with mpox will be enrolled in two clinics in remote settings in the DR Congo (Tunda and Kole general hospital) where mpox outbreaks are ongoing. After providing informed consent, participants will undergo standard ophthalmological examinations of their eyes to see if there are any complications of mpox. This includes history taking, clinical examination, technical examinations such as a dilated fundoscopic exam, a fluorescein test and a Schirmer test, and a conjunctival swab for tear collection for monkeypox virus (MPXV) detection. Pictures of the anterior and posterior segment will also be taken to aid later verification and interpretation of the study findings. If they are hospitalised for mpox (for clinical reasons or as part of their participation in another ongoing clinical trial at the study sites), they will be followed up for 14 days and examined during an unscheduled visit in the case of new or worsening severe issues. Otherwise, patients are followed up at day 14 (for those hospitalised), day 28 and day 59. Study participants will receive the same supportive eye care as non-study participants. Study participants will be compensated for their time lost and for transportation to the clinic.

The study will primarily assess the presence of ophthalmological signs and symptoms at enrollment, but also aims to describe the complications of mpox that may arise after that point in time.

ELIGIBILITY:
Inclusion Criteria:

* Patient of any age or gender with laboratory-confirmed infection with MPXV
* Laboratory confirmation of MPXV infection less than 48 hours before inclusion
* Patient or culturally acceptable representative is willing and able to give informed consent or assent for participation in the study

Exclusion Criteria:

* Patients for whom, in the judgment of the recruiting physician, participation in the study would interfere with routine optimal clinical care.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will take place in parallel to:
  * the PALM007 clinical trial (NCT05559099), which evaluates the efficacy of tecovirimat for the treatment of mpox in two sites in the Democratic Republic of the Congo: Tunda General Hospital, Maniema Province and Kole General Hospital, Sankuru Province.
  * The MBOTE study, which evaluates the clinical signs and symptoms in people with mpox at Kamituga General Hospital, South Kivu Province.
  Depending on the mpox epidemiological context other sites can be included at a later timepoint. The study may be continued after cessation of the PALM007 trial.
  Participants will be recruited among PCR-confirmed mpox cases, including but not limited to patients enrolled in the PALM 007 trial and MBOTE study. The study may be continued after cessation of the PALM007 trial and MBOTE study.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-29 (Estimated)

PRIMARY OUTCOMES:
Composite presence or absence of eye disease and visual deficiencies at presentation | At enrollment
  Composite presence of
  * orbital lesions (exophthalmos, enophthalmos, oculomotor paralysis...)
  * affection of the adnexa
  * affection of the anterior segment
  * affection of the posterior segment
  * affection of the optic nerve

SECONDARY OUTCOMES:
Ocular signs & symptoms at presentation and during follow-up | From enrollment until last follow-up
  Presence or absence of individual symptoms and signs over time
Visual acuity at presentation and during follow-up | From enrollment until last follow-up
  Result of Optotype letters/numbers and/or E test over time
presence of MPXV in tear fluid at presentation and during follow-up | From enrollment until last follow-up
  Result of MPXV-Polymerase Chain Reaction (PCR) on conjunctival swabs over time

CONTACTS AND LOCATIONS:
Overall Officials: Laurens Liesenborghs, Professor, Study Director — Institute of Tropical Medicine
Locations (1):
- Kamituga General Hospital, Kamituga, South Kivu, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Undecided